CLINICAL TRIAL: NCT00003395
Title: Dose-Ranging Study of Arsenic Trioxide in Advanced Hematologic Cancers
Brief Title: Arsenic Trioxide in Treating Patients With Advanced Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-023; CDR0000066395 (Registry Identifier: PDQ (Physician Data Query)); NCI-G98-1449
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; Waldenström macroglobulinemia; stage III multiple myeloma; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute eosinophilic leukemia; adult acute basophilic leukemia; adult acute megakaryoblastic leukemia (M7); progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; acute undifferentiated leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; adult acute monocytic leukemia (M5b); primary central nervous system non-Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; adult acute minimally differentiated myeloid leukemia (M0); intraocular lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; juvenile myelomonocytic leukemia; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Erythroblastic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Basophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Hairy Cell; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myelomonocytic, Juvenile; Lymphoma, B-Cell, Marginal Zone | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of arsenic trioxide in treating patients who have advanced hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Develop a safe, weight-based, extended-dosing regimen of arsenic trioxide suitable for outpatient therapy in patients with advanced hematologic cancers. II. Determine the pattern of clinical adverse experience in patients treated with this drug. III. Evaluate evidence of clinical responsiveness that may provide leads for further testing in patients treated with this drug.

OUTLINE: This is a dose-escalation study. Patients receive arsenic trioxide IV over 1-4 hours on days 1-25. Courses repeat every 3-5 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 4-6 patients receive escalating doses of arsenic trioxide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity. Patients are followed for 1 month.

PROJECTED ACCRUAL: Approximately 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven hematologic cancer, including acute or chronic leukemia, malignant lymphoma, or multiple myeloma Exclude acute promyelocytic leukemia (M3) Relapse from or resistance to at least one course of standard anticancer therapy and lack of alternative therapy that has proven to be curative in the underlying disease

PATIENT CHARACTERISTICS: Age: 17 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.5 mg/dL Renal: Creatinine no greater than 2.5 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception during and for at least 4 months after study No history of grand mal seizures (other than infantile febrile seizures) No active serious infections that are not controlled by antibiotics

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent cytotoxic chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: No other concurrent investigational agents

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-04; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Soignet, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States